CLINICAL TRIAL: NCT00587288
Title: An Efficacy and Safety Study of Reslizumab in the Treatment of Poorly Controlled Asthma in Subjects With Eosinophilic Airway Inflammation
Brief Title: Efficacy and Safety Study of Reslizumab to Treat Poorly Controlled Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ception Therapeutics (Industry)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Res-5-0010
Record Dates: First submitted 2008-01-04; First posted 2008-01-07 (Estimated); Results first posted 2016-04-26 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-07

CONDITIONS: Asthma
Keywords: Cinquil™; Reslizumab
MeSH Terms: conditions — Asthma | interventions — reslizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reslizumab 3 mg/kg (Experimental): Reslizumab 3 mg/kg intravenous (IV) on Day 0 of each 28-day (+/- 7 days) cycle, for 4 cycles
  Interventions: Biological: Reslizumab
- Placebo (Placebo Comparator): Saline placebo IV on Day 0 of each 28-day (+/- 7 days) cycle, for 4 cycles
  Interventions: Other: Saline

INTERVENTIONS:
Biological: Reslizumab
  Other Names: Cinquil™; CEP-38072; CTx55700
  Arms: Reslizumab 3 mg/kg
Other: Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of reslizumab in the treatment of subjects with poorly controlled asthma.

DETAILED DESCRIPTION:
Objectives:

Primary: To demonstrate the ability of reslizumab to improve asthma control in subjects with active asthma and eosinophilic airway inflammation.

Secondary:

* To study the ability of reslizumab to reduce induced sputum eosinophil (EOS) counts in subjects with asthma.
* To study the ability of reslizumab to reduce the number of eosinophilic clinical asthma exacerbations (CAE) in subjects with asthma. A CAE is defined as a ≥ 20% decrease in forced expiratory volume in 1 second (FEV1; absolute value) from the baseline value or a requirement for emergency treatment of asthma, hospital admission for asthma or treatment with three or more days of oral corticosteroids (OCS) for asthma worsening.
* To assess the safety and tolerability of reslizumab in subjects with asthma.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* male or female subjects aged ≥ 18 to 75 years at time of screening
* female if she is of non-childbearing potential, or of childbearing potential and willing to use specific barrier methods specified in protocol
* confirmation of asthma
* symptoms consistent with a diagnosis of asthma that is poorly controlled with an inhaled corticosteroid as determined by an Asthma Control Questionnaire (ACQ) score ≥ 1.5
* requirement for treatment with high dose daily fluticasone and at least one other agent for the treatment of asthma not specifically excluded in the protocol
* requirement for >/= 3% eosinophils in induced sputum at Screening

Exclusion Criteria:

* a clinically important event that would interfere with study schedule or procedure or compromise subject safety
* a diagnosis of hypereosinophilic syndrome
* an underlying lung disorder
* a current smoker
* use of systemic immunosuppressive agents within 6 months of study
* current use of systemic corticosteroids
* received attenuated live attenuated vaccines within three months prior to study entry
* expected to be poorly compliant with study drug, procedures, visits
* aggravating factors that are inadequately controlled
* participation in any investigational drug or device study within 30 days prior to study entry
* participation in biologics study within 3 months prior to study entry
* receipt of anti-human interleukin-5 (hIL-5) antibody within 6 months of study entry
* female subjects who are pregnant or nursing
* concurrent infection or disease that may preclude assessment of eosinophilic esophagitis
* concurrent immunodeficiency (human immunodeficiency [HIV], or acquired immunodeficiency syndrome [AIDS] or congenital immunodeficiency).
* current suspected drug and/or alcohol abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, MD, Study Director — Cephalon (Ception)
Locations (30):
- United States (24):
  - Children'S Hospital of Orange County-Pediatric Subspecialty Faculty, Orange, California
  - Allergy & Clinical Research Center, Centennial, Colorado
  - Asthma & Allergy Associates, P.C., Colorado Springs, Colorado
  - National Jewish Medical & Research Center, Denver, Colorado
  - Sneeze, Wheeze & Itch Associates, LLC, Normal, Illinois
  - Pulmonary Disease & Critical Care Associates, P.A., Columbia, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - Washington University of School of Medicine, St Louis, Missouri
  - The Asthma & Allergy Center, Papillion, Nebraska
  - Health Sciences Research at Asthma & Allergy, Cortland, New York
  - Wake Forest Univeristy Health Services, Winston-Salem, North Carolina
  - David Bernstein, Cincinnati, Ohio
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Clinical Research Institute of Southern Oregon, Medford, Oregon
  - Allergy and Asthma Specialists, Blue Bell, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Asthma Sinus Allergy Program & Research Centers, Nashville, Tennessee
  - Virginia Adult & Pediatric Allergy and Asthma, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Asthma, Inc, Seatle, Washington
  - Allergy, Asthma and Sinus Center, Greenfield, Wisconsin
  - University of Wisconsin-Madison, Allergy/Asthma Clinical Research Unit, Madison, Wisconsin
- Canada (6):
  - Heritage Medical Research Clinic, University of Calgary, Calgary, Alberta
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Queen's University, Richardson's House, Kingston, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Hopital du Sacre-Couer de Montreal, Montreal, Quebec
  - Hopital Laval, Québec, Quebec

REFERENCES:
- [Background] Castro M, Mathur S, Hargreave F, Boulet LP, Xie F, Young J, Wilkins HJ, Henkel T, Nair P; Res-5-0010 Study Group. Reslizumab for poorly controlled, eosinophilic asthma: a randomized, placebo-controlled study. Am J Respir Crit Care Med. 2011 Nov 15;184(10):1125-32. doi: 10.1164/rccm.201103-0396OC. Epub 2011 Aug 18. PMID 21852542

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reslizumab 3 mg/kg | Placebo
Started | 53 | 53
Completed | 50 | 44
Not Completed | 3 | 9
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 2 | 8
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Reslizumab 3 mg/kg: reslizumab 3 mg/kg IV on Day 0 of each 28-day (+/- 7 days) cycle, for 4 cycles
- Total: Total of all reporting groups
Arm/Group | Reslizumab 3 mg/kg | Placebo | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (13.94) | 45.8 (11.74) | 45.4 (12.83)
Age, Customized [Number; unit: participants]
  18 to < 45 years | 28 | 20 | 48
  45 to < 65 years | 19 | 32 | 51
  >/= 65 years | 6 | 1 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 29 | 63
  Male | 19 | 24 | 43

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to End of Therapy in Asthma Control Questionnaire (ACQ) Score
Description: The ACQ is a 7 question instrument. Each question has 7 possible answers of 0, 1, 2, 3, 4, 5, and 6. Each increasing value is an indication of poorer asthma control. At protocol specified visits, the participant answered questions 1 to 6, circling the response that best described how that participant was during the past week, on the basis of a daily diary for the week before the visit. At the actual visit, study center personnel reviewed the questions and responses with the participant and determined the response and score for question 7. The overall ACQ score was presented as the mean of these 7 individual scores and was a number between 0 and 6, but not necessarily an integer.
Time Frame: Baseline through End of Therapy (up to 15 weeks)
Population: Intent-to-treat (ITT) Analysis Set: all participants who received any amount of randomly assigned study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Reslizumab 3 mg/kg | Placebo
Number analyzed (Participants) | 53 | 53
units on a scale | -0.7 (1.02) | -0.3 (1.01)
Statistical Analysis 1: Comparison: Reslizumab 3 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.0541, ANCOVA — The p-value for the treatment comparison is based on the ANCOVA with adjustment for stratification factor and for variable at baseline; Adjusted mean difference = -0.38, 95% CI 2-sided [-0.76 to 0.01], Standard Error of Mean 0.194

2. Secondary Outcome: Percentage of ACQ Responders at End of Therapy
Description: Responders were defined as participants achieving at least a 0.5 reduction from baseline to End of Therapy in ACQ score. The ACQ is a 7 question instrument. Each question has 7 possible answers of 0, 1, 2, 3, 4, 5, and 6. Each increasing value is an indication of poorer asthma control. At protocol specified visits, the participant answered questions 1 to 6, circling the response that best described how that participant was during the past week, on the basis of a daily diary for the week before the visit. At the actual visit, study center personnel reviewed the questions and responses with the participant and determined the response and score for question 7. The overall ACQ score was presented as the mean of these 7 individual scores and was a number between 0 and 6, but not necessarily an integer.
Time Frame: Baseline, End of Therapy (up to 15 weeks)
Population: ITT Analysis Set: all participants who received any amount of randomly assigned study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Reslizumab 3 mg/kg | Placebo
Number analyzed (Participants) | 53 | 53
percentage of participants
  Responder = yes | 55 | 36
  Responder = no | 45 | 64
Statistical Analysis 1: Comparison: Reslizumab 3 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.0848, Regression, Logistic — The p-value for the treatment comparison was based on logistic regression with adjustment for stratification factor; Odds Ratio (OR) = 2.01, 95% CI 2-sided [0.91 to 4.46]

3. Secondary Outcome: Change From Baseline to End of Therapy in Forced Expiratory Volume in the First Second (FEV1)
Description: The change in FEV1 from baseline to End of Therapy was determined. FEV1 was measured during pulmonary function tests using standard spirometry measurements.
Time Frame: Baseline, End of Therapy (up to 15 weeks)
Population: ITT Analysis Set: all participants who received any amount of randomly assigned study drug with an assessment at Baseline and End of Therapy.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Reslizumab 3 mg/kg | Placebo
Number analyzed (Participants) | 52 | 52
L | 0.18 (0.372) | -0.08 (0.413)
Statistical Analysis 1: Comparison: Reslizumab 3 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.0023, ANCOVA — The p-value for the treatment comparison was based on the ANCOVA with adjustment for stratification factor and for variable at baseline; Adjusted mean difference = 0.240, 95% CI 2-sided [0.088 to 0.392], Standard Error of Mean 0.077

4. Secondary Outcome: Change From Baseline to End of Therapy in Percent Predicted FEV1
Description: The change in percent predicted FEV1 from baseline to End of Therapy was calculated from the FEV1 measured during pulmonary function tests using standard spirometry measurements. Each participant's percent predicted FEV1 was calculated by adjusting the FEV1 for age, sex, height and race. The percent predicted FEV1 was then calculated by comparing the predicted FEV1 to the observed FEV1 using the Crapo formula (Crapo et al 1981a, Crapo and Morris 1981b, Crapo et al 1982).
Time Frame: Baseline, End of Therapy (up to 15 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent predicted FEV1
Arm/Group | Reslizumab 3 mg/kg | Placebo
Number analyzed (Participants) | 52 | 52
percent predicted FEV1 | 6.2 (11.76) | -2.4 (12.93)
Statistical Analysis 1: Comparison: Reslizumab 3 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.0010, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Adjusted mean difference = 7.98, 95% CI 2-sided [3.30 to 12.65], Standard Error of Mean 2.36

5. Secondary Outcome: Mean Change From Baseline to End of Therapy in Induced Sputum Eosinophil Levels
Time Frame: End of Screening or Baseline, End of Therapy (up to 15 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change in eosinophil levels
Arm/Group | Reslizumab 3 mg/kg | Placebo
Number analyzed (Participants) | 38 | 36
percent change in eosinophil levels | -82.0 (66.88) | 45.9 (265.79)
Statistical Analysis 1: Comparison: Reslizumab 3 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.0068, ANCOVA — The p-value for the treatment comparison was based on the ANCOVA with adjustment for stratification factor and for variable at baseline. The difference between reslizumab 3.0 mg/kg and placebo groups was from comparison of the least square means; Adjusted mean difference = -125.29, 95% CI 2-sided [-214.81 to -35.77], Standard Error of Mean 44.885

6. Secondary Outcome: Percentage of Participants With Clinical Asthma Exacerbations (CAEs)
Description: A CAE was defined as a 20% or more decrease in forced expiratory volume in 1 second (FEV1, absolute value) from the baseline value, a requirement for emergency treatment of asthma, hospital admission for asthma, or treatment with 3 or more days of oral corticosteroids for asthma worsening.
Time Frame: up to 15 weeks
Population: ITT Analysis Set: all participants who received any amount of randomly assigned study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Reslizumab 3 mg/kg | Placebo
Number analyzed (Participants) | 53 | 53
percentage of participants | 8 | 19
Statistical Analysis 1: Comparison: Reslizumab 3 mg/kg vs Placebo; Test type: Superiority or Other; p = 0.0833, Regression, Logistic — The p-value for the treatment comparison was based on logistic regression with adjustment for stratification factor; Odds Ratio (OR) = 0.33, 95% CI 2-sided [0.10 to 1.15]
Statistical Analysis 2: Comparison: Reslizumab 3 mg/kg vs Placebo; Kaplan-Meier estimate of time to first CAE. (First quartile, median and third quartile "survival" times with 95% confidence intervals (ie, time to first CAE) could not be estimated since the proportion of patients experiencing CAE was too low. Therefore, the only number presented in regard to the Kaplan-Meier analysis is the p-value of the log-rank test, below. ); Test type: Superiority or Other; p = 0.0809, Log Rank; The p value for the treatment comparison was based on log rank test adjusting for stratification factor (ie, ACQ score ≤2 and >2)

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs), Serious AEs, and AEs Leading to Study Discontinuation
Description: Participants may have been included in more than 1 category. AEs summarized were those that began or worsened after dispensation of the study drug and before 30 days after the last dose of study drug. If the severity of an AE was missing, the AE was reported as "severe." If drug relationship of an AE was missing, the AE was reported as "probably related." WFT=withdrawn from treatment.
Time Frame: From start of study drug through 15 weeks + 30 days
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Reslizumab 3 mg/kg | Placebo
Number analyzed (Participants) | 53 | 53
participants
  Any AE | 38 | 42
  Severe or life-threatening AE | 3 | 1
  Treatment-related AE | 12 | 8
  Deaths | 0 | 0
  Serious AEs other than death | 2 | 1
  Treatment-related serious AEs | 0 | 0
  WFT or study due to AEs | 1 | 1
  WFT or study due to treatment-related AEs | 0 | 1

ADVERSE EVENTS:
Time Frame: From start of study drug through 15 weeks + 30 days
Arm/Group | Reslizumab 3 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/53 | 1/53
Other Adverse Events (participants affected / at risk) | 17/53 | 17/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reslizumab 3 mg/kg (N=53) | Placebo (N=53)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reslizumab 3 mg/kg (N=53) | Placebo (N=53)
FATIGUE (General disorders) | 4 (4) | 2 (2)
BRONCHITIS (Infections and infestations) | 2 (2) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 11 (14) | 5 (6)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (3) | 5 (5)
HEADACHE (Nervous system disorders) | 2 (3) | 5 (5)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.